CLINICAL TRIAL: NCT03911115
Title: Study of Food Preferences After Bariatric Surgery
Brief Title: Food Preferences After Bariatric Surgery (BariaTaste 3)
Acronym: BariaTaste3
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0219; 2019-A00774-53 (Other: ID-RCB)
Record Dates: First submitted 2019-04-05; First posted 2019-04-10 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric surgery: Individuals that have undergone a gastric bypass (RYGB) or a sleeve gastrectomy (SG)
  Interventions: Other: Food preference questionnaire

INTERVENTIONS:
Other: Food preference questionnaire — This is an online questionnaire administrated once to the participants, to assess food preferences after bariatric surgery. The investigating team will also collect data on the type of surgery, anthropometry, nutrition, taste, smell, disgust and intolerance as well as sociodemographic data.

SUMMARY:
Bariatric surgery is currently considered the most effective treatment for achieving significant, sustained weight loss and reducing comorbidities associated with obesity. Every year in France, more than 55,000 undergo this surgery and nearly 450 000 French have a history of surgery for obesity. The mechanisms of action of bariatric surgery are multiple and are not limited to caloric restriction. Neuro-hormonal effects, changes in the anatomy of the digestive tract, vagal changes or bile circulation have been identified as contributing factors to weight loss and postoperative improvement of comorbidities. In addition, post-operative changes in dietary preferences have also been described, which could contribute to initial weight loss and its maintenance over time (aversion to lipid and sugar products).

The counterpart of the rapid and durable efficacy of bariatric surgery is the exposure of patients to a significant risk of protein-energy malnutrition. It should be noted that the protein intake, very limited in the first months after surgery, remains well below the recommended intake after the first postoperative year. Spontaneous consumption of meat and vegetable protein is significantly reduced during the first postoperative month and up to one year after surgery. Apart from the limitation of gastric volume induced by surgery, clinical experience indicates that many patients turn away from protein consumption by aversion. A parallel was made between the significant drop in protein consumption during the first months and the initial loss of lean mass. Thus changes in dietary preferences induced by bariatric surgery could also contribute to postoperative nutritional risk (protein aversion).

At the same time, it is noted that olfactory and taste modifications have been reported in previous studies that could be associated with these changes in food preferences.

The hypotheses of the current study are that the type of surgery may affect dietary preferences differently after obesity surgery and that surgical failure may be associated with preferences for high fat, high sweet and low protein foods postoperatively for both types of surgery.

As far as the investigating team is aware, no study compares dietary preferences between sleeve gastrectomy and gastric bypass using this approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have undergone a Roux-en-Y Gastric Bypass (RYGB) or a sleeve gastrectomy (SG)
* Patient aged at least 18

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a bariatric surgery, Roux-en-Y Gastric Bypass (RYGB) or sleeve gastrectomy (SG)
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Food preferences | Day 0
  Food preferences will be measured using liking score for different food groups.The outcome will be assessed in the period following the bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Guyot, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France